CLINICAL TRIAL: NCT02181101
Title: Simultaneous Study of Gemcitabine-Docetaxel Combination Adjuvant Treatment, as Well as Extended Bisphosphonate and Surveillance-Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Collaborators: AstraZeneca (Industry); Chugai Pharma USA (Industry); Eli Lilly and Company (Industry); Novartis (Industry); Sanofi (Industry); Janssen Diagnostics, LLC (Industry)
Responsible Party: Principal Investigator, Prof. Dr. med. Harald Leo Sommer, Prof. Dr. med. Harald Leo Sommer, Ludwig-Maximilians - University of Munich
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SUCCESS-A; 2005-000490-21 (EudraCT Number)
Record Dates: First submitted 2014-06-04; First posted 2014-07-03 (Estimated); Last update posted 2014-07-03 (Estimated); Status verified 2014-07

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- AA-BA (Experimental): FEC-DocGemzar adjuvant chemotherapy; zoledronic acid i.v. 5 years
  Interventions: Drug: FEC-DocGemzar adjuvant chemotherapy; Drug: Zoledronic acid i.v. 5 years
- AB-BA (Experimental): FEC-Doc adjuvant chemotherapy; zoledronic acid i.v. 5 years
  Interventions: Drug: FEC-Doc adjuvant chemotherapy; Drug: Zoledronic acid i.v. 5 years
- AA-BB (Experimental): FEC-DocGemzar adjuvant chemotherapy; zoledronic acid i.v. 2 years
  Interventions: Drug: FEC-DocGemzar adjuvant chemotherapy; Drug: Zoledronic acid i.v. 2 years
- AB-BB (Active Comparator): FEC-Doc adjuvant chemotherapy; zoledronic acid i.v. 2 years
  Interventions: Drug: FEC-Doc adjuvant chemotherapy; Drug: Zoledronic acid i.v. 2 years

INTERVENTIONS:
Drug: FEC-DocGemzar adjuvant chemotherapy
  Arms: AA-BA; AA-BB
Drug: FEC-Doc adjuvant chemotherapy
  Arms: AB-BA; AB-BB
Drug: Zoledronic acid i.v. 2 years
  Arms: AA-BB; AB-BB
Drug: Zoledronic acid i.v. 5 years
  Arms: AA-BA; AB-BA

SUMMARY:
This is an open-label, multicenter, 2x2 factorial design, randomized controlled, Phase III study comparing the disease free survival after randomisation in patients treated with 3 cycles of Epirubicin-Fluorouracil-Cyclophosphamide(FEC)-chemotherapy, followed by 3 cycles of Docetaxel(Doc)-chemotherapy versus 3 cycles of Epirubicin-Fluorouracil-Cyclophosphamide(FEC), followed by 3 cycles of Gemcitabine-Docetaxel(DocGemzar)-chemotherapy, and to compare the disease free survival after randomisation in patients treated with 2 years of Zoledronate versus 5 years of Zoledronate in patients with early primary breast cancer. Patients will be required to have histopathological proof of axillary lymph node metastases (pN1-3) or high risk node negative, defined as: 'pT≥2 or histopathological grade 3, or age ≤ 35 or negative hormone receptor', but are not allowed to have evidence of distant disease. Patients will have to be entered into the study no later than 6 weeks after complete resection of the primary tumor. No other antineoplastic treatment other than surgical treatment, the defined cytotoxic and endocrine treatment and radiotherapy will be allowed prior to study entry and during the course of the study.

After surgery, leading to R0 resection of the invasive and intraductal components of the primary tumor, patients will be randomized to one of the following treatments:

First randomization

AA: 3 cycles of 5-Fluorouracil 500 mg/m² i.v. body surface area and Epirubicin 100 mg/m² i.v. and Cyclophosphamide 500 mg/m² i.v., (FEC100), each administered on day 1, repeated on day 22, subsequently followed by 3 cycles of Docetaxel 75 mg/m² body surface area i.v. (Doc), and Gemcitabine 1000 mg/m² i.v. (30 min infusion) (Gemzar), administered on day 1, followed by Gemcitabine 1000 mg/m² i.v. (30 min infusion) on day 8, repeated on day 22

AB: 3 cycles of 5-Fluorouracil 500 mg/m² i.v. body surface area and Epirubicin 100 mg/m² i.v. and Cyclophosphamide 500 mg/m² i.v., (FEC100), each administered on day 1, repeated on day 22, subsequently followed by 3 cycles of Docetaxel 100 mg/m² body surface area i.v. (Doc), administered on day 1, repeated on day 22

Second randomization B

BA: Zoledronic acid 4 mg i.v., every 3 months for the duration of two years, subsequently followed by zoledronic acid 4 mg i.v., every 6 months for the duration of additional three years

BB: Zoledronic acid 4 mg i.v., every 3 months for the duration of two years

During the zoledronic acid treatment period, patients will receive 500 mg Calcium p.o. qid and 400 i.E. Vitamin D p.o. qid.

Patients with positive hormone receptor status (≥ 10 % positively stained cells for estrogen and/or progesterone) of the primary tumor will receive Tamoxifen treatment 20 mg p.o. per day for 2 years, after the end of chemotherapy. Subsequent to chemotherapy, postmenopausal patients with positive hormone receptor status will be treated with Anastrozole (Arimidex®) 1 mg p.o. for additional 3 years, premenopausal patients will continue Tamoxifen treatment for additional 3 years. In addition to tamoxifen, all patients with positive hormone receptor status of the primary tumor and under the age of 40 or restart of menstrual bleeding within 6 months after the completion of cytostatic treatment or with premenopausal hormone levels as defined below will receive Goserelin (Zoladex®) 3.6 mg subcutaneously every 4 weeks over a period of 2 years following chemotherapy. Premenopausal endocrine status will be assumed, if the following serum levels are met: Luteinizing hormone (LH) < 20 mIE/ml, follicle stimulating hormone (FSH) < 20 mIE/ml and estradiol (E2) > 20 pg/ml. Endocrine therapy will start after the end of chemotherapy.

All patients with breast conserving therapy or more than 3 axillary lymph node metastases or in the following cases after mastectomy:

* T3/T4-carcinoma
* T2-carcinoma > 3 cm
* multicentric tumor growth
* lymphangiosis carcinomatosa or vessel involvement
* involvement of the pectoralis fascia or a safety margin < 5 mm.

will receive adjuvant radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Primary epithelial invasive carcinoma of the breast pT1-4, pM0
* Histopathological proof of axillary lymph node metastases (pN1-3) or high risk pN0/NX, defined as: 'pT ≥ 2 or histopathological grade 3 or age ≤ 35 or negative hormone receptor status'
* Complete resection the primary tumor with margins of resection free of invasive carcinoma not more than 6 weeks ago
* Females ≥ 18 years of age
* Performance Status ≤ 2 on Eastern Cooperative Oncology Group (ECOG) Scale
* Adequate bone marrow reserve: leucocytes ≥ 3.0 x 10^9/l and platelets ≥ 100 x 10^9/l
* Bilirubin within one fold of the reference laboratory's normal range, aspartate aminotransferase (ASAT) (serum glutamate oxalacetate transaminase, SGOT), alanine aminotransferase (ALAT) (serum glutamate pyruvate transaminase, SGPT) and alkaline phosphatase (AP) within 1,5 fold of the reference laboratory's normal range for patients
* Intention of regular follow-up visits for the duration of the study
* Ability to understand the nature of the study and to give written informed consent

Exclusion Criteria:

* Inflammatory breast cancer
* Previous or concomitant cytotoxic or other systemic antineoplastic treatment which is not part of or allowed within this study
* History of treatment or disease affecting bone metabolism (e.g., Paget's disease, primary hyperparathyroidism)
* Prior treatment with bisphosphonates within the last 6 months
* Severe renal insufficiency as evidenced by creatinine clearance < 30 ml/min as calculated using the Cockcroft-Gault formula
* Second primary malignancy (except in situ carcinoma of the cervix or adequately treated basal cell carcinoma of the skin)
* Cardiomyopathy with impaired ventricular function (New York Heart Association Functional Classification Class (NYHA) > II), cardiac arrythmias influencing left ventricular ejection fraction (LVEF) and requiring medication, history of myocardial infarction or angina pectoris within the last 6 months, or arterial hypertension not being controlled by medication
* Any known hypersensitivity against docetaxel, epirubicin, cyclophosphamide, fluorouracil, gemcitabine or any other medication included in the study protocol
* Use of any investigational agent within 3 weeks prior to inclusion
* Patients in pregnancy or breast feeding (in premenopausal women anticonception has to be assured: intra uterine devices, surgical methods of sterilization, or, in hormone unsensitive tumors only, oral, subcutaneous or transvaginal hormonal, non estrogen containing contraceptives)
* Current active dental problems including infection of the teeth or jawbone (maxilla or mandibular); dental or fixture trauma, or a current or prior diagnosis of osteonecrosis of the jaw (ONJ), of exposed bone in the mouth, or of slow healing after dental procedures.
* Recent (within 6 weeks) or planned dental or jaw surgery (e.g.. extraction, implants)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3754 (Actual)
Dates: Start 2005-09; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Disease free survival | 5 years

SECONDARY OUTCOMES:
Overall survival | 5 years
Number of adverse events related to cancer therapy observed | 5 years
Quality of life | 5 years
  Changes in quality of life over time as defined by EORTC QLQ-C30 and QLQ-BR23 questionnaire
Number of skeletal/bone-related adverse events observed including osteonecrosis of the jaw | 5 years
Number of patients who develop malignant disease other than recurrence of the breast cancer treated within the trial | 5 years
Distant disease free survival | 5 years
  Disease free survival excluding ipsilateral breast tumor recurrence, regional invasive recurrences, contralateral breast cancer, and all in situ carcinomas

CONTACTS AND LOCATIONS:
Overall Officials: Harald L Sommer, Prof. Dr. med., Study Director — Ludwig-Maximilians - University of Munich
Locations (1):
- Klinikum der Universität München, Klinik und Poliklinik für Frauenheilkunde und Geburtshilfe, Campus Innenstadt, Munich, Bavaria, Germany

REFERENCES:
- [Derived] Friedl TWP, Fehm T, Muller V, Lichtenegger W, Blohmer J, Lorenz R, Forstbauer H, Fink V, Bekes I, Huober J, Juckstock J, Schneeweiss A, Tesch H, Mahner S, Brucker SY, Heinrich G, Haberle L, Fasching PA, Beckmann MW, Coleman RE, Janni W, Rack B. Prognosis of Patients With Early Breast Cancer Receiving 5 Years vs 2 Years of Adjuvant Bisphosphonate Treatment: A Phase 3 Randomized Clinical Trial. JAMA Oncol. 2021 Aug 1;7(8):1149-1157. doi: 10.1001/jamaoncol.2021.1854. PMID 34165508
- [Derived] de Gregorio A, Haberle L, Fasching PA, Muller V, Schrader I, Lorenz R, Forstbauer H, Friedl TWP, Bauer E, de Gregorio N, Deniz M, Fink V, Bekes I, Andergassen U, Schneeweiss A, Tesch H, Mahner S, Brucker SY, Blohmer JU, Fehm TN, Heinrich G, Lato K, Beckmann MW, Rack B, Janni W. Gemcitabine as adjuvant chemotherapy in patients with high-risk early breast cancer-results from the randomized phase III SUCCESS-A trial. Breast Cancer Res. 2020 Oct 23;22(1):111. doi: 10.1186/s13058-020-01348-w. PMID 33097092
- [Derived] Deniz M, DeGregorio A, DeGregorio N, Bekes I, Widschwendter P, Schochter F, Ernst K, Scholz C, Bauer EC, Aivazova-Fuchs V, Weissenbacher T, Kost B, Jueckstock J, Andergassen U, Steidl J, Trapp E, Fasching PA, Haberle L, Beckmann MW, Schneeweiss A, Schrader I, Janni W, Rack B, Friedl TW. Differential prognostic relevance of patho-anatomical factors among different tumor-biological subsets of breast cancer: Results from the adjuvant SUCCESS A study. Breast. 2019 Apr;44:81-89. doi: 10.1016/j.breast.2018.12.008. Epub 2018 Dec 20. PMID 30690254
- [Derived] Vilsmaier T, Rack B, Janni W, Jeschke U, Weissenbacher T; SUCCESS Study Group. Angiogenic cytokines and their influence on circulating tumour cells in sera of patients with the primary diagnosis of breast cancer before treatment. BMC Cancer. 2016 Jul 27;16:547. doi: 10.1186/s12885-016-2612-7. PMID 27464822
- [Derived] Jueckstock J, Rack B, Friedl TW, Scholz C, Steidl J, Trapp E, Tesch H, Forstbauer H, Lorenz R, Rezai M, Haberle L, Alunni-Fabbroni M, Schneeweiss A, Beckmann MW, Lichtenegger W, Fasching PA, Pantel K, Janni W; SUCCESS Study Group. Detection of circulating tumor cells using manually performed immunocytochemistry (MICC) does not correlate with outcome in patients with early breast cancer - Results of the German SUCCESS-A- trial. BMC Cancer. 2016 Jul 7;16:401. doi: 10.1186/s12885-016-2454-3. PMID 27387743
- [Derived] Widschwendter P, Friedl TW, Schwentner L, DeGregorio N, Jaeger B, Schramm A, Bekes I, Deniz M, Lato K, Weissenbacher T, Kost B, Andergassen U, Jueckstock J, Neugebauer J, Trapp E, Fasching PA, Beckmann MW, Schneeweiss A, Schrader I, Rack B, Janni W, Scholz C. The influence of obesity on survival in early, high-risk breast cancer: results from the randomized SUCCESS A trial. Breast Cancer Res. 2015 Sep 18;17(1):129. doi: 10.1186/s13058-015-0639-3. PMID 26385214
- See also: Related Info — http://success-studie.de/